CLINICAL TRIAL: NCT04634643
Title: Pathophysiologic Mechanisms Leading to Intrahepatic Fat Accumulation in Obese Youth
Brief Title: Pathogenesis of Pediatric Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000028731; R01MD015974 (NIH)
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Usual diet and physical activity — Patients will be followed up to assess the effect of the usual diet and physical activity on development of NAFLD

SUMMARY:
The main aim of the study is to discover the mechanisms underlying the pathophysiology of NAFLD in obese youth.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common hepatic disease in pediatrics, affecting about 30% of obese youth. The term NAFLD defines a wide spectrum of disease severity ranging from simple intrahepatic fat accumulation without liver injury (steatosis) to nonalcoholic steatohepatitis (NASH), fibrosis and cirrhosis.

A 20-year retrospective study has shown that subjects who develop NAFLD during their youth have about 13 times higher mortality rate for end-stage liver disease than healthy subjects of similar age and gender. NAFLD is highly prevalent among Hispanic youth, while non-Hispanic Black (NHB) youth are protected against intrahepatic fat accumulation even in the presence of severe obesity and insulin resistance. Understanding the pathophysiology underlying these differences could shed new light on the mechanisms leading to NAFLD in obese youth.

Preliminary data suggest that Hispanic and NHB obese youth might have a different ability to metabolize carbohydrates (CHO) through glycolysis, with Hispanics showing higher glycolysis than NHB. Therefore, Hispanics might experience a higher rated tricyclic acid cycle (TCA) and hepatic de novo lipogenesis (DNL).

In the present study, the investigators aim to address the following questions:

1. Is the different susceptibility between Hispanics and NHB in developing NAFLD due to a higher capability of Hispanics to metabolize CHO through glycolysis, TCA cycle and DNL?
2. Do these metabolic changes anticipate the onset of the disease in Hispanic youth?
3. Are the higher rates of glycolysis, TCA and DNL driven by high but not pathologic changes in glucose levels over time?

To address these aims, the investigators plan to recruit 30 Hispanics and 30 NHB obese youth and to measure glycolysis by using a new method to assess lactate kinetics and to determine the TCA cycle and DNL by using 13C-Propionate and D2O.

The investigators will also assess glycolysis and intrahepatic fat content in a group of 200Hispanic obese youth without fatty liver at baseline every 12 months for two years to determine whether higher glycolytic rates precede intrahepatic fat accumulation. To assess whether metabolic changes in glycolysis are driven by higher but not-pathologic glucose levels, the investigators will measure glucose changes over ten days every six months by using a continuous glucose monitoring system. If successful, these studies will provide novel insight into the pathogenesis of pediatric NAFLD and will open new avenues to test novel therapeutic approaches.

Study was paused in 2022 and reopened recruitment in November 2023.

ELIGIBILITY:
Inclusion Criteria:

* Good general health, taking no medication on a chronic basis;
* age 12 to 18 years, in puberty (girls and boys: Tanner stage II-V);
* BMI >85th for obese cohort;

Exclusion Criteria:

* Baseline creatinine >1.0 mg; pregnancy;
* the presence of endocrinopathies (e.g. Cushing syndrome);
* cardiac or pulmonary or other significant chronic illness;
* adolescents with a psychiatric disorder or with substance abuse;
* monogenic obesity syndromes;
* use of drugs affecting intrahepatic fat content (e.g.; liraglutide, fish oil, etc.).

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Hispanics and NHB youth with and without NAFLD
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Lactate synthesis | 60 months
  lactate synthesis will be measured during an oral glucose tolerance test by measuring lactate. Synthetic rates will be measured by using a mathematical model.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Santoro, MD, PhD, Principal Investigator — Associate Professor of Pediatrics (Endocrinology)
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT04634643/ICF_000.pdf